CLINICAL TRIAL: NCT00400452
Title: Manual Wheelchair Skills Training for Long-term-care Residents: A Pilot Randomized Controlled Trial of Efficacy
Brief Title: Manual Wheelchair Skills Training for Long-term-care Residents
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: poor enrollment
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Cher Smith, Capital District Health Authority, Canada
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: CDHA014
Record Dates: First submitted 2006-11-15; First posted 2006-11-16 (Estimated); Last update posted 2011-07-06 (Estimated); Status verified 2009-07

CONDITIONS: Healthy; Wheelchair Users
Keywords: wheelchair; skills; long-term-care; caregivers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: wheelchair skills training

SUMMARY:
It is hypothesized that, compared to a control group, manual wheelchair users and their caregivers in the long-term-care setting who receive the wheelchair skills training program will improve their wheelchair skills to a statistically significant extent and will retain these improvements for at least one month.

ELIGIBILITY:
Inclusion Criteria (wheelchair user):

* be seventeen (17) or older
* be a manual wheelchair user, living in a long-term-care facility;
* be expected to require the long-term use of a wheelchair (at least four [4] hours/week for at least eight [8] weeks), as reported by a clinical therapist;
* be competent to give informed consent (as indicated by a Mini Mental State Examination score of 20 or higher) or have a proxy with power of attorney willing to provide consent,
* have the verbal endorsement of the clinical therapist (if any) to participate;
* have the written permission of the attending physician to participate;
* be willing to take part in the study, including signing the consent after carefully reading it.

Exclusion Criteria (wheelchair user):

* have an unstable medical condition (e.g. angina, seizures), as determined by the attending physician, house staff or ERN;
* have an emotional or psychiatric problem of a type or extent that might make participation unpleasant, as determined by the attending physician, house staff or ERN.

Inclusion Criteria (caregiver):

* be seventeen (17) or older;
* provide at least part-time [at least one (1) hour/week] wheelchair-handling care for a wheelchair user in a long-term-care facility;
* be willing to take part in the study, including signing the consent form after carefully reading it.

Exclusion Criteria (caregiver):

* have an unstable medical condition (e.g. angina, seizures), as indicated by self-report;
* have an emotional or psychiatric problem of a type or extent that might make participation unpleasant, as indicated by self-report.

Min Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2007-05; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Wheelchair Skills Test

SECONDARY OUTCOMES:
demographics
Mini-Mental State Examination score

CONTACTS AND LOCATIONS:
Overall Officials: Cher Smith, Principal Investigator — Capital Health, Department of Occupational Therapy
Locations (1):
- Camp Hill Veteran's Memorial Building, Capital Health, Halifax, Nova Scotia, Canada

REFERENCES:
- [Result] Smith C, Kirby RL. Manual wheelchair skills capacity and safety of residents of a long-term-care facility. Arch Phys Med Rehabil. 2011 Apr;92(4):663-9. doi: 10.1016/j.apmr.2010.11.024. Epub 2011 Mar 2. PMID 21367398
- See also: Related Info — http://www.wheelchairskillsprogram.ca